CLINICAL TRIAL: NCT06829212
Title: A Prospective Clinical Trial to Evaluate the Safety and Efficacy of Implantable Wireless Recording System (WRS) for General Control of External Devices in Paralyzed/Amputee Patients
Brief Title: Research on Wireless Brain Implant System for General Control of External Devices
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai StairMed Technology Co., Ltd. (Industry)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2302-CL-01-001; 2024-1325 (Other: Huashan Hospital Institutional Review Board)
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Complete or Incomplete Paraplegia/quadriplegia; Spinal Cord Injury; Brainstem Stroke; Amyotrophic Lateral Sclerosis; Bilateral Upper Limb Amputation
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries; Brain Stem Infarctions; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implantation (Experimental): Implantation of the WRS64
  Interventions: Device: WRS

INTERVENTIONS:
Device: WRS — WRS is a minimally invasive, wireless brain-machine interface system, consisting of a wireless implanted neural signal collector(Model: WRS64), data energy transmitter(Model: DTC01/02), and a brain function information management platform software(Model: SW01).

SUMMARY:
The clinical trial aims to evaluate the safety and efficacy of the minimally invasive, wireless brain-machine interface system (WRS) in enabling general brain control of external devices, such as a cursor and other assistive technologies, for paralyzed and amputee patients.

WRS integrates a high-throughput, ultra-flexible neural electrode with an extremely small cross-sectional size-approximately one-hundredth the diameter of a human hair. Moreover, the implantable component is fully embedded within the body, leaving no visible external traces.

DETAILED DESCRIPTION:
The investigators' technology is designed to assist paralyzed and amputee patients in regaining certain physical functions, thereby improving participants' overall quality of life and daily convenience.

The investigators hope to enable participants to achieve general control over external devices through neural signals in this clinical trial. This eliminates the need for manual manipulation to control devices such as a cursor or other assistive technologies, which can be operated solely through thought. Such advancements will facilitate enhanced communication with loved ones, support the acquisition of new skills, and provide more accessible opportunities for entertainment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years (inclusive), any gender.
* Diagnosed with spinal cord injury, brainstem stroke, amyotrophic lateral sclerosis, or other motor neuron diseases causing partial or complete paralysis, or bilateral upper limb amputation.
* Diagnosis stable for at least 6 months before screening, with the condition present for at least 1 year.
* Willing to follow the study protocol and attend all visits, with or without caregiver assistance.
* Informed consent signed by participant and/or caregiver, with full understanding of the trial's purpose.

Exclusion Criteria:

* Previous implantation of metal objects or devices (except dental implants or non-impacting implants).
* Long-term use of anticoagulants/antiplatelets with insufficient cessation, or abnormal coagulation test results.
* Unable to tolerate anesthesia or surgery.
* Severe neurological disorders or brain injury leading to significant dysfunction.
* Scalp conditions that may impair wound healing.
* Acute or severe infections.
* Cognitive impairment or psychiatric disorders.
* Severe dysfunction of vital organs, malignancies, or autoimmune diseases.
* Life expectancy under 1 year.
* Drug or alcohol abuse.
* Pregnant, breastfeeding, or planning pregnancy during the study.
* Other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Device-Related Adverse Events (AE) | Through study completion, an average of 7 months

SECONDARY OUTCOMES:
Adverse Events | Through study completion, an average of 7 months
Serious Adverse Event | Through study completion, an average of 7 months
BPS | At an average of 4 to 7 months after implantation, both before and during the follow-up phases.
  Bits per second, determined by the net number of correct targets selected per minute (NTPM) during task participation by the subject, and the grid size.
Usage Time (hours/month) | At an average of 5 to 7 months after implantation, during the follow-up phases.
  The amount of time the subject uses the experimental device each month.
Accuracy | At an average of 5 to 7 months after implantation, during the follow-up phases.
  The percentage of correctly completed commands from the total commands in the predefined task list, which are independently completed by the subject within a specified time.
Psychological State | At an average of 4 to 7 months after implantation, both before and during the follow-up phases.
  The subject and/or their caregiver will complete the checklist to assess psychological states and other relevant indicators (each question is graded from 1 to 5, with lower values being better).
Caregiver Burden | At an average of 4 to 7 months after implantation, both before and during the follow-up phases.
  The subject's caregiver will complete the checklist to assess caregiver burden and other related indicators (each question is scored from 0 to 4, with lower scores being better).

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No